CLINICAL TRIAL: NCT03016988
Title: Bortezomib Combined With Fludarabine and Cytarabine for Mantle Cell Lymphoma Patients：a Single Arm, Open-labelled, Phase 2 Study
Brief Title: The Efficacy and Safety of Bortezomib Combined With Fludarabine and Cytarabine Treatment for Mantle Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tingbo Liu (Other)
Collaborators: Union hospital of Fujian Medical University (Other)
Responsible Party: Sponsor-Investigator, Tingbo Liu, Professor of medicine, Fujian Medical University
Organization: Fujian Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fujian Medical University
Record Dates: First submitted 2016-10-11; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-08

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Bortezomib; Fludarabine; Cytarabine
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bortezomib; fludarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib,Fludarabine and Cytarabine (Other): Bortezomib(V) 1.3mg/m2, subcutaneously,day 1,4,8,11; Fludarabine(F) 25mg/m2, intravenously day 1-3; Cytarabine(A) 500mg/m2 for 3 days(day1-3).
  Interventions: Drug: Bortezomib; Drug: Fludarabine; Drug: Cytarabine

INTERVENTIONS:
Drug: Bortezomib — Bortezomib(V) 1.3mg/m2, subcutaneously,day 1,4,8,11;
  Other Names: Bortezomib (PS-341)
Drug: Fludarabine — Fludarabine(F) 25mg/m2, intravenously day 1-3;
  Other Names: NSC 118218
Drug: Cytarabine — Cytarabine(A) 500mg/m2 for 3 days(day1-3)
  Other Names: Cytosar-U; Cytosine Arabinoside

SUMMARY:
Mantle cell lymphoma (MCL) is a type of non-Hodgkin's lymphoma (NHL) and shows poor survival. This study to evaluate the efficacy and safety of Bortezomib combined with Fludarabine and Cytarabine treatment in the naive and relapsed MCL who are not eligible for high dose therapy and transplantation.

DETAILED DESCRIPTION:
The eligibility criteria were pathologically confirmed, previously untreated MCL or relapsed MCL as defined by the World Health Organization classification; age≥18 years; Eastern Cooperative Oncology Group (ECOG) performance status of 0-2; adequate haematologic function (haemoglobin > 9.0 g/l, absolute neutrophil count > 1500/ml, platelets > 75,000/l), hepatic function (total serum bilirubin ≤ 1.5 times the upper limit of normal, alanine aminotransferase and aspartate aminotransferase ≤ 2.5 times the upper limit of normal), renal function (serum creatinine ≤ 1.5 mg/dl, creatinine clearance ≥ 50 ml/min); normal coagulation function and electrocardiogram results. Stage was defined according to the Ann Arbor system.

The Fujian Medical University Union Hospital approved this study before subjects were enrolled.

Treatment dosages were as follows:

days 1,4,8,and 11 subcutaneous infusion of 1.3mg/m2 Bortezomib. Days 1-3 intravenous infusion 25mg/m2 Fludarabine. Days 1-3 intravenous infusion of 500mg/m2 Cytarabine. The regimen was repeated every 28 days for a maximum of six cycles.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. pathologically confirmed, previously untreated MCL or relapsed MCL as defined by the World Health Organization classification;
2. age≥18 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
4. adequate haematologic function (haemoglobin > 9.0 g/l, absolute neutrophil count > 1500/ml, platelets > 75,000/l),
5. adequate hepatic function (total serum bilirubin ≤ 1.5 times the upper limit of normal, alanine aminotransferase and aspartate aminotransferase ≤ 2.5 times the upper limit of normal),
6. adequate renal function (serum creatinine ≤ 1.5 mg/dl, creatinine clearance ≥ 50 ml/min);
7. normal coagulation function and electrocardiogram results.
8. willingness to provide written informed consent.

Exclusion Criteria:

1. MCL patients who do NOT response or are refractory to preview treatment.
2. Who do NOT sign the consent form.
3. whose life expectation is less than 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | Follow-up to 36 months
  Interval from registration to progression or death from any cause

SECONDARY OUTCOMES:
Overall response rate | Up to 36 months
  Lugano classification

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Cheah CY, Seymour JF, Wang ML. Mantle Cell Lymphoma. J Clin Oncol. 2016 Apr 10;34(11):1256-69. doi: 10.1200/JCO.2015.63.5904. Epub 2016 Jan 11. PMID 26755518